CLINICAL TRIAL: NCT07008417
Title: A Single-center, Randomized, Open-label, Two-formulation, Two-cycle, Two-sequence, Single-dose, Crossover Bioequivalence Study of Cabergoline Tablets Under Fasting and Postprandial Conditions in Healthy Chinese Subjects
Brief Title: A Study on Bioequivalence of Cabergoline Tablets in Human Body
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GenSci127-101
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Hyperprolactinemia
MeSH Terms: conditions — Hyperprolactinemia | interventions — Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cabergoline tablets test formulation (Experimental): Administration order: Cabergoline test formulation(T), Cabergoline reference formulation(R)
  Interventions: Drug: Cabergoline tablets test formulation
- Cabergoline tablets reference formulation (Experimental): Administration order: Cabergoline reference formulation(R), Cabergoline test formulation(T)
  Interventions: Drug: Cabergoline tablets reference formulation

INTERVENTIONS:
Drug: Cabergoline tablets test formulation — Single oral administration
  Arms: Cabergoline tablets test formulation
Drug: Cabergoline tablets reference formulation — Single oral administration
  Arms: Cabergoline tablets reference formulation

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of the test formulation and reference formulation of cabergoline tablets in healthy Chinese subjects under fasting and postprandial conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18-45 years (including boundary values), male or female;
* Body mass index: 19-26 kg/m2 (including boundary values), male weight ≥50 kg, female weight ≥45 kg;
* Normal results of physical examination, vital signs, laboratory tests, 12 lead-ECG, chest X-ray, abdominal ultrasound, or non-clinical significance changes in the assessments above.

Exclusion Criteria:

* Received camergoline treatment within the past six months; Those who have a history of allergy to carergoline or any drug component; Those who have had a history of allergy to two or more drugs, foods, etc.
* Those who currently have the following clinically significant diseases, including but not limited to peripheral vascular lesions, orthostatic hypotension, valvular heart disease, fibrous lesions, severe peptic ulcers and other diseases, or have a previous history of related diseases; Or those with other related diseases of the respiratory system, circulatory system, digestive system, blood system, endocrine system, immune system, skin system, mental and nervous system, otorhinolaryngology, etc., which have been judged by researchers as having clinical significance;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-05-06 (Estimated)

PRIMARY OUTCOMES:
Cmax | : 0 hours-72 hours post-administration
AUC0-72h | 0 hours-72 hours post-administration

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang, China